CLINICAL TRIAL: NCT01699035
Title: Survivor Perspective on Critical Factors to Return to Work After Stroke
Brief Title: Survey on Return to Work After Stroke
Status: Completed | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Hartke, Lead Psychologist, Shirley Ryan AbilityLab
Other Study IDs: H133B080031
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: stroke; work; vocational rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke survivors: stroke survivors who have either returned to work, have thought about returning to work, or have tried to return to work

SUMMARY:
Survey of survivor perspective on critical elements that either facilitate or inhibit return to work after a stroke. Critical elements are queried in areas of finances, stroke impairments, interpersonal support, therapeutic support, organization influences, work or job specific issues and psychological issues.

DETAILED DESCRIPTION:
The objective of this project is to more accurately describe the stroke survivor's perspective on return to work. The survey development included qualitative analysis of a set of interviews with stroke survivors to arrive at the critical elements described above, followed by item development with an expert panel and preliminary testing of the wording and format for legibility. The survey is being administered both on-line and by paper through the mail to a wide range of survivors with the objective of obtaining a large, diverse sample. The ultimate goal of the project is to arrive at a refined set of recommendations to inform stroke survivors, health care professionals and employers to increase their sensitivity to the needs and desires of individual attempting to return to work after stroke.

ELIGIBILITY:
Inclusion Criteria:

* have returned to work, have thought about returning to work, or have tried to return to work

Exclusion Criteria:

* non-stroke disability
* retired or no plan to return to work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke survivors
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
critical factors that facilitate or inhibit return to work after stroke | after collection of data on all surveys
  38 multiple choice items that assess psychological factors important to return to work, financial incentives and disincentives, the role of stroke impairments, interpersonal supports that facilitate and inhibit return, the role of therapeutic support especially vocational rehabilitation, organizational influences, and work specific issues that impact on return. Demographic information is also queried including work type and current work status. Data will be analyzed descriptively by these critical factors and also by other demographic factors such as age, work status, and race.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hartke, Ph.D., Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Hartke RJ, Trierweiler R, Bode R. Critical factors related to return to work after stroke: a qualitative study. Top Stroke Rehabil. 2011 Jul-Aug;18(4):341-51. doi: 10.1310/tsr1804-341. PMID 21914598